CLINICAL TRIAL: NCT02929394
Title: Maintenance Therapy With Trabectedin Versus Observation After First Line Treatment With Doxorubicin of Patients With Advanced or Metastatic Soft Tissue Sarcoma.
Brief Title: Trabectedin Maintenance Post 1st-line in STS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1447-STBSG; 2016-003535-38 (EudraCT Number)
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2019-11

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Histologically proven locally advanced or metastatic high grade STS (excluding histologies insensitive to chemotherapy such as ASPS, PECOMA subtypes)
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational treatment (Active Comparator): Trabectedin 1.2 mg/m² through a central venous catheter as an IV infusion over 24 hours every 4 weeks until disease progression (RECIST 1.1) or unacceptable toxicity.
  Interventions: Drug: Trabectedin
- observation (No Intervention): Observation through clinical and radiological follow-up until disease progression (RECIST 1.1).

INTERVENTIONS:
Drug: Trabectedin — Trabectedin 1.2 mg/m² through a central venous catheter as an IV infusion over 24 hours every 4 weeks until disease progression (RECIST 1.1) or unacceptable toxicity
  Other Names: Yondelis
  Arms: investigational treatment

SUMMARY:
Maintenance therapy with trabectedin versus observation after first line treatment with doxorubicin of patients with advanced or metastatic soft tissue sarcoma.

This is a prospective, multicenter, randomized, open label Phase III trial investigating whether a maintenance treatment with trabectedin, as compared to the observational approach, can prolong progression-free survival in patients with advanced, inoperable and/or metastatic STS after response or stabilisation during first line treatment with doxorubicin.

DETAILED DESCRIPTION:
Progression free survival will be estimated by the Kaplan-Meier method. The median survival time and its associated 95% non-parametric CI will be provided. Rates at 3 month intervals will be estimated using the log-log transformation of the Kaplan-Meier estimates and the standard deviation of the Kaplan Meier estimate based on the Greenwood formula.

For the primary analysis, PFS from randomization will be compared between the two arms using the score test from a Cox proportional hazards model adjusted for histology (stratification factor). The corresponding estimate of the treatment effect (hazard ratio) and 95% CI will be provided.

Secondary analyses include:

* the primary comparison of PFS repeated using methods for interval-censored data to adjust for deviations from the planned imaging scheduled, if any.
* the above mentioned analyses performed for PFS measured from date of starting firstline doxorubicin treatment.

Overall survival and time to second progression (PFS2) measured from randomization and from starting firstline doxorubicin treatment will be estimated by the Kaplan-Meier method. The median times and their associated 95% non-parametric CI will be calculated. Rates at 3 month intervals will be estimated using the log-log transformation of the Kaplan-Meier estimates and the standard deviation of the Kaplan Meier estimate based on the Greenwood formula. They will be compared between the two arms using an adjusted Cox proportional hazards model; the corresponding estimates of the hazard ratio and 95% CI will be provided. The above mentioned PFS2 comparison will also be repeated using methods for interval-censored data.

The adverse events related to the treatment (excluding those declared not reasonably possibly related to the treatment, but including those with relationship not assessable) will be described in the safety population. Worst grade of the AEs will be tabulated. Whenever a CTCAE code exists, the grade will be displayed according to that system, otherwise the values will be coded in up to three categories as below lower limit of normal (LLN), within normal range, and above upper limit of normal (ULN), as deemed appropriate.

The percentage of patients presenting severe treatment-related AE (grade ≥ 3), of patients reported to have died of toxicity and of patients who stopped treatment due to toxicity will be calculated and the 95% confidence interval will be presented.

ELIGIBILITY:
* Histologically proven locally advanced or metastatic high grade STS (excluding histologies insensitive to chemotherapy such as ASPS, PECOMA subtypes)
* Non-progressive disease (CR, PR or SD according to RECIST 1.1) after 6 cycles of first-line chemotherapy with doxorubicin for advanced and/or metastatic malignant STS.
* Interval from last dose of doxorubicin to start of treatment is maximum 6 weeks.
* Prior neoadjuvant or adjuvant non-anthracycline-chemotherapy is allowed, provided that the disease did not progress during neoadjuvant and/or adjuvant therapy or within 12 weeks after completion of the perioperative treatment.
* Representative formalin fixed, paraffin embedded tumor blocks or 10 unstained tissue slides, either from the primary tumor or a metastatic lesion, must be available for histological central review. Histological central review is not required before treatment start but it is mandatory to send unstained tumor slides (blocks optional) at time of study entry. Local histopathological diagnosis will be accepted for entry into this trial.

Age 18 years or older WHO performance status ≤ 1

Adequate bone marrow, liver and renal function and coagulation parameters:

* neutrophils ≥ 1.5 x 109/L;
* hemoglobin ≥ 9 g/dL (or ≥ 5.6 mmol/L). Blood transfusions or the administration of hematopoietic growth factors are allowed to achieve these baseline values;
* platelets ≥ 100 x 109/L;
* Total bilirubin ≤ ULN;
* Albumin > 30g/L
* SGPT/ALT and SGOT/AST ≤ 2.5 x ULN for patients with liver metastasis or patients with Gilbert syndrome bilirubin ≤ ULN;
* Creatine phosphokinase (CPK) ≤ 2.5 x ULN;
* Alkaline phosphatase ≤ 2.5 x ULN (consider hepatic isoenzymes 5-nucleotidase or gamma glutamyl transpeptidase (GGT), if the elevation could be osseous in origin); Creatinine clearance/eGFR >30mL/minmin as per local standard method
* Normal cardiac function (LVEF assessed by MUGA or ECHO within normal range of the institution), normal 12 lead ECG (without clinically significant abnormalities). The following unstable cardiac conditions are not allowed:
* Congestive heart failure
* Angina pectoris
* Myocardial infarction within 1 year before registration/randomization
* Uncontrolled arterial hypertension defined as blood pressure ≥ 150/100 mm Hg despite optimal medical therapy
* Arrhythmias clinically significant
* No prior exposure to trabectedin
* Recovery from toxicity (no more than Grade 1, except for alopecia)
* No active or uncontrolled infections or serious illnesses or medical conditions, including a history of chronic alcohol abuse, hepatitis, HIV and/or cirrhosis.
* No active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy is allowed if administered as stable dose for at least one month before randomization)
* No history, within the past five years, of malignancies other than soft tissue sarcoma (except: basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, resected incidental prostate cancer staged pT2 with Gleason Score 6 and postoperative PSA < 0.5 ng/ml). Patients with any history of malignancies who are disease-free for more than 5 years are eligible.
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 3 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female patients who are breast feeding should discontinue nursing prior to the first dose of study treatment.and until 3 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Important note: All eligibility criteria must be adhered to, in case of deviation discussion with Headquarters and study coordinator is mandatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
progression-free survival | until 3/4 years after randomization of the first patient
  The primary end-point is progression-free survival defined from randomization according to RECIST 1.1.

SECONDARY OUTCOMES:
Safety and tolerability (Common Toxicity Criteria CTCAE 4.0) | until 3/4 years after randomization of the first patient
Overall survival | until 3/4 years after randomization of the first patient
Time to second progression (PFS2) | until 3/4 years after randomization of the first patient
Health related quality of life (QLQ-C30) | until 3/4 years after randomization of the first patient

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gelderblom, Study Chair — Leiden University Medical Centre
Locations (14):
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Assistance Publique - Hopitaux de Marseille - Hôpital de La Timone, Marseille
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover
  - UniversitaetsMedizin Mannheim, Mannheim
- Leiden University Medical Center, Leiden, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Spain (3):
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Barcelona
  - Hospital Universitario San Carlos, Madrid
- Royal Marsden Hospital - Chelsea, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All publications must comply with the terms specified in the EORTC Policy 009 "Release of Results and Publication Policy".